CLINICAL TRIAL: NCT02460185
Title: The Role of Maternal Physical Exercise on Spontaneous Labor Onset - A Randomized Clinical Trial
Brief Title: Role of Maternal Physical Exercise on Spontaneous Labor Onset
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Lisboa Norte (Other)
Responsible Party: Principal Investigator, Isabel Pereira, M.D., Centro Hospitalar Lisboa Norte
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MPEX
Record Dates: First submitted 2015-05-29; First posted 2015-06-02 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy; Labour Onset and Length Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Without maternal physical exercise practice
- Study Group (Active Comparator): Behavioral: 30 minutes of walking, 3 times a week at 4 Km/h. Induction of labor was performed at 41 weeks.
  Interventions: Behavioral: Study group: Maternal Physical Exercise

INTERVENTIONS:
Behavioral: Study group: Maternal Physical Exercise — Exercise: 30 minutes of walking, 3 times a week at 4 Km/h.
  Arms: Study Group

SUMMARY:
Evaluate the effects of the practice of maternal physical exercise on the term of pregnancy as a method to enhance spontaneous labor.

DETAILED DESCRIPTION:
At 38 weeks low-risk pregnant women, with singleton cephalic fetus and without previous cesarean delivery, were randomized into 2 groups: a control group without maternal physical exercise practice and a study group with 30 minutes of walking, 3 times a week at 4 Km/h. Induction of labor was performed at 41 weeks

ELIGIBILITY:
Inclusion Criteria:

* 38 weeks low-risk pregnant women
* singleton cephalic fetus
* without previous cesarean delivery

Exclusion Criteria:

* pathological pregnancy
* twin pregnancy
* previous cesarean section

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Rate of labor induction | 41 weeks
  Rate of labor induction will be analysed

SECONDARY OUTCOMES:
Gestational age on spontaneous labor onset | 5 week
  Gestational age will be analysed on spontaneous labor onset
Active stage duration | 1 day
Cesarean section rate | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Barros Pereira, M.D., Principal Investigator — Departamento de Obstetricia, Ginecologia e Medicina da Reprodução, Centro Hospitalar Lisboa Norte, Hospital de Santa Maria
Locations (1):
- Departamento de Obstetricia, Ginecologia e Medicina da Reprodução, Lisbon, Portugal

REFERENCES:
- [Derived] Pereira IB, Silva R, Ayres-de-Campos D, Clode N. Physical exercise at term for enhancing the spontaneous onset of labor: a randomized clinical trial. J Matern Fetal Neonatal Med. 2022 Feb;35(4):775-779. doi: 10.1080/14767058.2020.1732341. Epub 2020 Mar 29. PMID 32223479